CLINICAL TRIAL: NCT00439491
Title: Role of Adipose Tissue in Pathogenesis of Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 303040158
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2007-02-23 (Estimated); Status verified 2007-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin resistance; Hypocaloric diet; Adipose tissue; adipocytokine
MeSH Terms: conditions — Obesity; Insulin Resistance

INTERVENTIONS:
Behavioral: Hypocaloric diet

SUMMARY:
The aim of the study was to investigate the relationship between insulin resistance and body composition in relation to secterion and expression of adipocytokines. Obese subjects undergo 6 months hypocaloric diet and, before, during and at the end of the diet, plasma samples and subcutaneous adipose tissue samples are obtained for subsequent analysis. In addition, body composition and insulin resistance are measured before and during the diet.

DETAILED DESCRIPTION:
The aim of the study was to investigate the relationship between insulin resistance and body composition in relation to secterion and expression of adipocytokines. Obese subjects undergo 6 months hypocaloric diet without any medication and, before, during and at the end of the diet, plasma samples and subcutaneous adipose tissue samples are obtained for subsequent analysis. Adipose tissue samples are obtained using needle biopsy. In addition, before and during the diet,body composition is measured using multifrequency bioimpedance and insulin resistance is evaluated using either hyperinsulinemic clamp or glucose/insulin - derived indices.

ELIGIBILITY:
Inclusion Criteria:

* Obesity

Exclusion Criteria:

* Diabetes
* Coronary heart disease
* Eating disorders
* Medication of beta blockers
* Medication of antiobesity drugs

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35
Dates: Start 2004-01; Study Completion 2006-12

PRIMARY OUTCOMES:
Body weight
Body fat

SECONDARY OUTCOMES:
Insulin resistance
Adipocytokine plasma levels
Adipocytokine adipose tissue expression

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Stich, Ass Prof MD PhD, Principal Investigator — Third Faculty of Medicine, Charles Uniersity in Prague
Locations (1):
- Third Faculty of Medicine, Charles University in Prague, Prague, Czechia

REFERENCES:
- See also: web page of the Third Faculty of Medicine — http://www.lf3.cuni.cz